CLINICAL TRIAL: NCT06681532
Title: Bovine Pericardium Membrane Versus Native Collagen Membrane in Conjunction With Sticky Bone Graft in Treatment of Class II Furcation Defects in Lower Molars: A Randomized Controlled Trial.
Brief Title: Bovine Pericardium Membrane Versus Native Collagen Membrane in Conjunction With Sticky Bone Graft in Treatment of Class II Furcation Defects in Lower Molars.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibrahim Ahmed Zein Elabdin Ahmed (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Ahmed Zein Elabdin Ahmed, BDS, Principal Investigator, Oral Medicine, and Periodontology Department., Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A05030240M
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Are treated with open flap debridement, native collagen membrane and bovine bone graft particles.
  Interventions: Procedure: Native collagen membrane and bovine bone graft in treatment of class II furcation defects in lower molars
- Study group (Experimental): Are treated with open flap debridement, bovine pericardium membrane and bovine bone graft particles.
  Interventions: Procedure: Bovine pericardium membrane and bovine bone graft in treatment of class II furcation defects in lower molars

INTERVENTIONS:
Procedure: Native collagen membrane and bovine bone graft in treatment of class II furcation defects in lower molars — The bovine bone graft particles will be mixed with concentrated growth factor (CGF) to form sticky bone, the furcation defect area will be condensed with the mixture and covered completely with native collagen membrane.
  Arms: Control group
Procedure: Bovine pericardium membrane and bovine bone graft in treatment of class II furcation defects in lower molars — the bovine bone graft particles will be mixed with concentrated growth factor (CGF) to form sticky bone, the furcation defect area will be condensed with the mixture and covered completely with bovine pericardium membrane.
  Arms: Study group

SUMMARY:
Materials and methods: Twenty five patients (n=25) were selected from the outpatient clinic of the department of oral medicine and periodontology at Mansoura university's faculty of dentistry, 5 patients (n=5) were excluded as they didn't meet the inclusion criteria or met one or more of the exclusion criteria.

The participants 20 patients exhibiting one buccal or lingual mandibular molar furcation defect were assigned into two treatment groups: group I (control group), group II (study group), 10 patients in each group.

Patients in group I will be treated with open flap debridement, native collagen membrane and bovine bone graft particles. Patients in group II will be treated with open flap debridement, bovine pericardium membrane and bovine bone graft particles.

Periodontal assessment (plaque index (PI), gingival index (GI), horizontal clinical attachment level (HCAL), vertical clinical attachment level (VCAL), gingival recession (REC) and probing depth (PD)) will be evaluated at baseline, 3 months and 6 months after periodontal treatment.

Radiographic assessment using CBCT (bone loss in the horizontal direction (BL-H), bone loss in vertical direction (BL-V), length of the root trunk (RT), width of furcation entrance (FW) will be evaluated at baseline and 6 months after periodontal treatment.

DETAILED DESCRIPTION:
Study population:

The randomized controlled clinical trial includes 20 participants selected from the outpatient clinic of the department of oral medicine and periodontology at Mansoura university's faculty of dentistry from July 2024 to September 2024. All the patients exhibits one buccal or lingual mandibular molar furcation defect.

Study Design:

A double blinded, parallel group randomized controlled trial. The participants were randomly assigned using a computer random number generator program into two treatment groups:

* Group 1: The control group, includes 10 patients with class II furcation defects in lower molars and will be treated with open flap debridement, native collagen membrane and bovine bone graft particles.
* Group 2: The study group, includes 10 patients with class II furcation defects in lower molars and will be treated with open flap debridement, bovine pericardium membrane and bovine bone graft particles.

Surgical procedure:

Two weeks prior to surgery, using ultrasonic scaler tips and micro curettes, the remaining periodontal pocket will be treated. Only the exposed root surface and the first 3 mm of the root beneath the periodontal pocket will be instrumented. In order to guarantee proper manipulation, surgery won't start until the marginal tissue has a fibrous tone and there is little to no inflammation.

Following injection of local anesthetic (articaine/epinephrine 1:100,000), sulcular incisions will be made, a full thickness flap will be elevated at the furcation site, extending at least one tooth mesial and distal to the affected tooth, and extending beyond mucogingival junction for adequate accessibility. Furcation micro curettes and ultrasonic scalers will be used to fully debride and clean the furcation area, and then the area will be carefully irrigated with saline.

After this, In (Group 1&2), the bovine bone graft particles will be mixed with concentrated growth factor (CGF) to form sticky bone, the defect area will be condensed with the mixture and covered completely with native collagen membrane (group 1) or bovine pericardium membrane (group 2), both will be trimmed, adapted and placed so as to completely cover the grafted area and the adjacent 2-3 mm of bone tissue. Bioabsorbable ligatures will be used to secure the membrane to the soft tissues adjacent to the site of regeneration, preventing graft movement and membrane collapse. Afterwards, the flaps will be repositioned and securely sutured.

All patients will be prescribed amoxicillin 500 mg every 8 hours for duration of 5 days (azithromycin 500 mg once daily for 3 days for patients allergic to amoxicillin). Postoperative pain and inflammation will be managed with ibuprofen 600 mg (or acetaminophen 1g for patients allergic to ibuprofen). Patients will be instructed to rinse with 0.2% chlorhexidine twice daily for one week, without engaging in mechanical hygiene in the surgical area. Sutures will be removed after one week, and patients will be advised to perform mechanical cleaning of the area using a soft brush and apicocoronal brushing.

Follow-up visits will be scheduled at 1, 2, 3, and 4 weeks to assess patient-reported feedback, adherence to postoperative instructions and , clinical examination (Parameters such as bleeding, swelling, discomfort -eating and speech-, and pain are evaluated), as well as at 3 and 6 months, also incorporating supportive periodontal therapy and reinforcement of oral hygiene practices.

Periodontal assessment:

The clinical assessment will be performed at baseline, 3 months and 6 months after periodontal treatment.

1. Probing depth (PD), measured from the free gingival margin to the bottom of the sulcus.
2. Horizontal clinical attachment level (HCAL) is measured with Naber's probe measure the depth of FI.
3. Vertical clinical attachment level (VCAL), measured using UNC-15 probe from cemento-enamel junction to the bottom of the sulcus.
4. Gingival recession (REC), measured on the buccal aspect, at the level of the central axis of the tooth, from the CEJ to the gingival margin.
5. Plaque index (PI), introduced by Silness and Loe in 1964.
6. Gingival Index (GI), developed by Loe and Silness in 1963.

Radiographic assessment:

Radiographic interpretation of the furcation defect will be done using CBCT small field of view of the operated site taken for hard tissue assessment, at baseline and 6 months post-operatively.

The three axes (axial, sagittal, and coronal) of the CBCT images will be analyzed continuously. The linear measurements of the dimension of bone loss in the horizontal and vertical directions (BL-H, BL-V), root trunk (RT), and furcation width (FW) will be assessed.

* Bone loss in the horizontal direction (BL-H): using the axial view to measure the distance between the outer root surface and the inter- radicular bone, measured to the nearest millimeter.
* Vertical bone loss (BL-V): using the sagittal view to measure the distance from the furcation entrance (FE) to the base of the defect (BD) in the vertical direction.
* Length of the root trunk (RT): using the sagittal view to measure the distance from the cementoenamel junction (CEJ) to the furcation entrance (FE).
* Width of furcation entrance (FW): using the axial or sagittal view to measure the widest mesial-distal distance in the furcation.

This study is conducted following guidelines regulating research work on human subjects of the Faculty of Dentistry, Mansoura University, and the study protocol was reviewed and approved by the Research Ethics Committee of the Faculty of Dentistry, Mansoura University, Egypt. (Number: A05030240M)

Sample size calculation was based on efficacy of using a bovine pericardium membrane with a bovine bone graft versus a native collagen membrane with bovine bone graft for treatment of class II furcation defects, retrieved from previous research ( Serroni et al., 2022). Using G power program version 3.1.9.7 to calculate sample size based on effect size of 0.816 ,using 2-tailed test , α error =0.05 and power = 90.0% , the total calculated sample size will be 8 in each group at least .

Pretreatment period, Patients receive detailed information about their treatment, including potential effects, risks, and alternative options. The patients must have a broad understanding of this explanation and be legally competent to provide written consent before any necessary procedures.

Statistical Assessment:

Data will be analyzed using statistical package for social sciences (SPSS) version 22. Qualitative data will be presented as number and percent, Quantitative data will be tested for normality by Shapiro-Wilk test then described as mean and standard deviation for normally distributed data and median and range for non-normally distributed. The appropriate statistical test will be applied according to data type with the following suggested tests: Chi-Square for categorical variable, Spearman or Pearson correlation will be used to correlate continuous variables. : Kruskal Wallis test and One Way ANOVA test for non-normally and normally distributed data for more than 2 independent groups.

ELIGIBILITY:
Inclusion criteria:

* Display a buccal or lingual class II furcation defect (Hamp et al. classification) in their lower molars.
* The tooth with a horizontal clinical attachment level (HCAL) greater than 3mm and a probing depth (PD) greater than or equal to 6mm in the mid-buccal or mid-lingual sites.
* Have not undergone any periodontal treatment in the past 6 months.
* A plaque index score (PI) below 1 at surgery, assessed using the Ramfjord teeth.

Exclusion Criteria:

* Patients with class I or class III furcation defects.
* Systemic disease contraindicating periodontal surgery.
* Taking any medication that may have an impact on their periodontal health within the last 6 months.
* Smoking.
* Being pregnant or lactating.
* Teeth with periapical lesions and teeth with mobility.
* Third molars or teeth with improper endodontic or restorative treatment.
* Patients with furcation caries, metal crowns in the furcation area or amalgam fillings near the alveolar crest.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical ( Horizontal clinical attachment level [HCAL] ) | 6 months
  Is measured with Naber's probe, measure the depth of Furcation.
Radiographic ( Bone loss in the horizontal direction [BL-H] ) | 6 months
  Using the CBCT axial view to measure the distance between the outer root surface and the inter-radicular bone.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim A Zein Elabdin, Principal Investigator — Mansoura university Faculty of dentistry
Locations (1):
- Faculty of dentistry , Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided